CLINICAL TRIAL: NCT05918159
Title: Effects of Sarcopenia on the Fall Risk, Body Composition, General Health Status and Quality of Life in Elderly: a Population-based Study
Brief Title: Effects of Sarcopenia on General Health Status in Elderly: a Population-based Study
Status: Completed | Type: Observational
Sponsor: Universidade do Algarve (Other)
Collaborators: European Regional Development Fund (Other)
Responsible Party: Sponsor
Other Study IDs: 0348_CIE_6_E_2
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Sarcopenia; Sarcopenic Obesity; Frailty
Keywords: Sarcopenia; Quality of Life; Frailty; Muscle Strength; Aging; Body Composition; Postural Balance; Falls
MeSH Terms: conditions — Sarcopenia; Frailty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples were collected with the COBAS b 101 system and after analyzing by the system, the samples were immediately destroyed and deposited in waste suitable for biological residues.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly: Group of 274 elderly
  Interventions: Other: Sarcopenia Assessment

INTERVENTIONS:
Other: Sarcopenia Assessment — The prevalence of sarcopenia in a group of elderly people and its correlation with other health variables was determined.

SUMMARY:
This is a observational study, that aimed to determine the prevalence of sarcopenia using European Wording Group on Sarcopenia in Older People (EWGSOP) algorithm in a general elderly population in Algarve region (Portugal). Because muscle is metabolically active tissue, sarcopenia may also contribute to the development of some of the metabolic disorders associated with aging. However, the risk factors associated with sarcopenia are poorly understood. Thus, a cross-sectional survey of a sample of 274 elderly adults aged 60 or over, were included in the study. Correlations of sarcopenia with functional level, lipid and glycemic profile, nutritional and physical activity level, fall risk, quality of life, and self-reported comorbidities will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 60 years;
* Live in the community;
* Independet Gait.

Exclusion Criteria:

* Presence of moderate or severe cognitive impairment;
* Presence of uncontrolled cardiovascular disease and active cancer;
* Use of a pacemaker;
* Use of internal prosthesis.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants of this study are people from the community of the Algarve region over 60 years old.
  To proceed with the recruitment of participants, the study was disseminated through promotional materials, such as flyers and posters in senior universities, institutions/associations, municipalities and parish councils, sports complexes, among other community spaces in the Algarve region.
  A non-probabilistic sampling was used. The sampling process consisted in a first phase of intentional sampling, which allowed recruiting many individuals over 60 years old who met the inclusion and exclusion criteria and in a second phase the sampling process was also carried out using the snowball method.
Sampling Method: Non-Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Prevalence of Sarcopenia in elderly population | 0 Months
  Determine the prevalence of sarcopenia using European Wording Group on Sarcopenia in Older People (EWGSOP) algorithm in a general elderly population in Algarve region.
Quality of life in elderly population | 0 Months
  Quality of life was assessed at one time point only (due to the nature of the cross-sectional study design) using the subscore and total score of Medical Outcomes Study 36-item Short-Form Health Survey instrument. Instrument scores can range between 0 - 100. Higher values mean better self-perception of quality of life.

SECONDARY OUTCOMES:
Cognitive Assessment | 0 Months
  Cognitive Assessment was assessed by the instrument Montreal Cognitive Assessment (MoCA). Instrument with a maximum score of 30 points, where higher scores mean better cognitive performance.
Body mass index (kg/m2) - body composition | 0 Months
  Body mass index (kg/m2) was measured using the bioimpedance technique.
Fat Mass (kg and %) - body composition | 0 Months
  Fat Mass (kg and %) was measured using the bioimpedance technique.
Fat-Free Mass (kg and %) - body composition | 0 Months
  Fat-Free Mass (kg and %) was measured using the bioimpedance technique.
Fat Mass Index (kg/m2) - body composition | 0 Months
  Fat Mass Index (kg/m2) was measured using the bioimpedance technique.
Fat-Free Mass Index (kg/m2) - body composition | 0 Months
  Fat-Free Mass Index (kg/m2) was measured using the bioimpedance technique.
Muscle Mass Index (kg/m2) - body composition | 0 Months
  Muscle Mass Index (kg/m2) was measured using the bioimpedance technique.
Total body water (L and %) - body composition | 0 Months
  Total body water (L and %) was measured using the bioimpedance technique.
Resistence (Ohms) - body composition | 0 Months
  Resistence (Ohms) was measured using the bioimpedance technique.
Reactance (Ohms) - body composition | 0 Months
  Reactance (Ohms) was measured using the bioimpedance technique.
Phase angle (angle) - body composition | 0 Months
  Phase angle was measured using the bioimpedance technique.
Visceral fat (L) - body composition | 0 Months
  Visceral fat (L) was measured using the bioimpedance technique.
High-density lipoprotein (HDL) cholesterol (mg/dL) - Lipid Profile | 0 Months
  High-density lipoprotein (HDL) cholesterol (mg/dL) was measured taking a sample blood which was analysed by the COBAS b 101 system.
Low-density lipoprotein (LDL) cholesterol (mg/dL) - Lipid Profile | 0 Months
  Low-density lipoprotein (HDL) cholesterol (mg/dL) was measured taking a sample blood which was analysed by the COBAS b 101 system.
Triglycerides (mg/dL) - Lipid Profile | 0 Months
  Triglycerides (mg/dL) was measured taking a sample blood which was analysed by the COBAS b 101 system.
Total cholesterol (mg/dL) - Lipid Profile | 0 Months
  Total cholesterol (mg/dL) was measured taking a sample blood which was analysed by the COBAS b 101 system.
Glicemic Profile in elderly | 0 Months
  Glicemic Profile was measured by COBAS b 101 system, taking a sample blood which was analysed for Glycated Hemoglobin (HbA1c).
Inflammatory levels in elderly population | 0 Months
  Inflammatory levels was measured by COBAS b 101 system, taking a sample blood which was analysed for C-reactive protein - CRP.
Nutritional level in elderly population | 0 Months
  Nutrional level was assessed at one time point only (due to the nature of the cross-sectional study design) using a questionnaire Mini Nutritional Assessment. Instrument scores can range between 0 - 30. The cutoff points used were: 0-7 points - malnourished; 8-11 points - at risk of malnutrition; 12-24 points - normal nutritional status.
Postural Stability in elderly population | 0 Months
  Postural stability was assessed by a force platform using the length displacement of center of pressure.
Peak Torque (N/m) of Quadriceps and Hamstring Muscles | 0 Months
  Peak Torque of Quadriceps and Hamstring Muscles was measured by afixed dynamometer with concentric/concentric action at an angular velocity of 60º per second for 5 repetitions of extension and flexion of each knee.
Work (N/m) of Quadriceps and Hamstring Muscles | 0 Months
  Work of Quadriceps and Hamstring Muscles was measured by afixed dynamometer with concentric/concentric action at an angular velocity of 60º per second for 5 repetitions of extension and flexion of each knee.
Power (N/m) of Quadriceps and Hamstring Muscles | 0 Months
  Power of Quadriceps and Hamstring Muscles was measured by afixed dynamometer with concentric/concentric action at an angular velocity of 60º per second for 5 repetitions of extension and flexion of each knee.
Peak torque time (s) of Quadriceps and Hamstring Muscles | 0 Months
  Peak torque time of Quadriceps and Hamstring Muscles was measured by afixed dynamometer with concentric/concentric action at an angular velocity of 60º per second for 5 repetitions of extension and flexion of each knee.
Force (kg) of Quadriceps and Hamstring Muscles | 0 Months
  Force of Quadriceps and Hamstring Muscles was measured by afixed dynamometer with concentric/concentric action at an angular velocity of 60º per second for 5 repetitions of extension and flexion of each knee.
Time up and Go (TUG) test - Fall risk in elderly population | 0 Months
  TUG test measures (in seconds) the time a person needs to rise from a chair with armrests, to walk the distance of 3 m with usual assistive devices, if necessary, turn, return to the chair, and sit down. TUG test is a composite measure of functional mobility. It includes transfer tasks (standing up and sitting down), walking, and turning, thus incorporating neuromuscular components such as power, agility, and balance. Faster test completion signals better dexterity and functional state, whereas the score of ≥13.5 was used as a cut-off point to identify the elderly individuals who are at risk for falls in community dwelling.
Modified Falls Efficacy Scale (MFES) - Fall risk in elderly population | 0 Months
  The Modified Falls Efficacy Scale (MFES) consists of 14 items to be subjectively evaluated on a scale of 1 to 5 in terms of confidence in the ability of a person to perform daily indoor and outdoor activities without falling. Higher values represent less risk of falling.
Physical Activity level in elderly population | 0 Months
  Physical activity level was assessed at one time point only (due to the nature of the cross-sectional study design) using the questionnaire PASE - Physical Activity Scale for Elderly. The PASE measures the level of self-reported physical activity in individuals aged 65 years or older and is comprised of items regarding occupational, household, and leisure activities during the previous 7-day period. It was used frequency, duration, and intensity level of activity over the previous week to assign a score, ranging from 0 to 793, with higher scores indicating greater physical activity.
Pain associated with osteoarthritis | 0 Months
  Pain associated with osteoarthritis was mesured by Western Ontario and McMaster Universities Arthritis Index (WOMAC Index) - subscore pain. This instrument is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales: Pain (5 items), Stiffness (2 items), and Physical Function (17 items). The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Higher scores indicate worse pain, stiffness, and functional limitations.
Stiffness associated with osteoarthritis | 0 Months
  Pain associated with osteoarthritis was mesured by Western Ontario and McMaster Universities Arthritis Index (WOMAC Index) - subscore pain. This instrument is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales: Pain (5 items), Stiffness (2 items), and Physical Function (17 items). The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Higher scores indicate worse pain, stiffness, and functional limitations.
Physical Function associated with osteoarthritis | 0 Months
  Pain associated with osteoarthritis was mesured by Western Ontario and McMaster Universities Arthritis Index (WOMAC Index) - subscore pain. This instrument is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales: Pain (5 items), Stiffness (2 items), and Physical Function (17 items). The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Higher scores indicate worse pain, stiffness, and functional limitations.
Functional Level of Lower Limbs | 0 Months
  To assess the functionality of the lower limbs, the Lower Extremity Functional Scale (LEFS) instrument was applied. The lower extremity functional scale is a valid patient-rated outcome measure for the measurement of lower extremity function. The score can vary between 0 and 80, with higher values representing better functionality.
Handgrip strength (HGS) | 0 Months
  HGS was measured with the handgrip Dynamometer Lafayette Digital 5030D1 in both upper limbs.
Identifies the concerns and priorities of older people | 0 Months
  Following the World Health Organisation, the "Integrated care for older people" (ICOPE) guidelines, each assessment with Age Care Technologies (ACT) Assessment generates a report which lists identifies concerns and priorities for action, together with several summary scores to measure needs, risks and outcomes, including: Quality of life, Falls risk, Vision, Hearing, Activities of Daily Living, Nutrition, Locomotor, Oral Health, Accommodation, Finances, Cognition, Depression, Loneliness, Social participation, and Violence against older people.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra R Pais, PhD, Principal Investigator — Universidade do Algarve
Locations (1):
- Marta Botelho, Faro, Algarve, Portugal